CLINICAL TRIAL: NCT01848249
Title: Deceased Donor Urinary Biomarkers to Predict Kidney Transplant Outcomes
Brief Title: Deceased Donor Biomarkers and Recipient Outcomes
Acronym: DDS
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 1206010465; R01DK093770-01A1 (NIH)
Record Dates: First submitted 2013-04-30; First posted 2013-05-07 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Deceased Donor Kidney Transplant; Acute Kidney Injury; Delayed Graft Function; End Stage Renal Disease; Graft Failure
Keywords: deceased donors; kidney donor; transplant recipients; kidney transplant; delayed graft function; biomarkers; end stage renal disease; graft failure
MeSH Terms: conditions — Acute Kidney Injury; Delayed Graft Function; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ((A)) Urine Samples: At time of deceased donor nephrectomy ((B)) Perfusates: At time of initiation and stopping of machine perfusion
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Deceased-Donor Cohort: We will collect urine samples from approximately 1600 deceased donors and approximately 600 perfusate samples from machine-pumped kidneys from participating organ procurement organizations (OPOs).
- Recipient Cohort (Overall and Detailed): No samples will be collected from the recipients. Only clinical data and outcomes will be collected from the recipients.

SUMMARY:
Compared to chronic dialysis, kidney transplantation provides recipients with longer survival and better quality of life at a lower cost. In order to meet increasing demands for kidney allografts, kidneys from older and sicker donors are being procured. This has led to greater discard rates of donated kidneys as well as more complications for recipients, including shorter allograft survival. Available clinical models to predict kidney allograft quality have poor prognostic ability and do not asses the degree of kidney allograft injury. However, allograft injury near the time of procurement can lead to major consequences for the transplant recipient: greater risks of delayed graft function, poor allograft function and premature loss of the transplant. Our proposal is based on the hypotheses that novel biomarkers measured in donor urine and transport media at the time of procurement can assess acute and chronic kidney injury and that distinct biomarker patterns will predict allograft survival. In collaboration with five organ procurement organizations, we will collect urine samples from consecutive deceased donors and samples of transport solution for every pumped kidney. We will measure markers of injury, repair, inflammation and fibrosis. We will determine mortality and allograft survival in all patients by linkage to the United Network for Organ Sharing (UNOS) database (Overall Cohort). Additionally, we will perform a detailed chart review of a subset of recipients (detailed cohort) and will also examine associations between biomarkers and longitudinal graft function over five years after transplant. Early, non-invasive and rapid assessment of donor kidney injury could drive better allocation decisions and potentially reduce the rates of post-transplant complications. Further, these new tools could provide a platform for clinical trials of therapies for allografts and kidney transplant recipients aimed at ameliorating allograft injury.

DETAILED DESCRIPTION:
Our study has several key processes that we have developed and tested to address our scientific aims:

1. Enrollment

   We will collect urine samples from approximately 1600 deceased donors and approximately 600 perfusate samples from machine-pumped kidneys from participating organ procurement organizations (OPOs). We estimate that our final donor group will be comprised of 55% standard criteria donors, 25% expanded-criteria donors and 10% donors after cardiac death. Approximately, 20% of the kidneys will be discarded.
2. Donor Data

   Donor variables come from two sources: the United Network for Organ Sharing (UNOS) database and detailed data abstraction from each OPO. The UNOS database provides data on all donors with demographics and other important clinical characteristics. The additional data collected by the OPO staff captures granular information on events surrounding donor death, which are not included in the UNOS database. These data will be available on all enrolled donors and include variables such as serial serum creatinine, nadir blood pressures, medication and vasopressor use, and machine pump parameters.
3. Overall Recipient Cohort

   Over 2000 recipients will have received kidneys from the deceased donors in our study. The Overall Cohort will comprise all of these recipients General demographic and clinical characteristics about recipients in the Overall Cohort will come from the UNOS database. For the Overall Recipient Cohort, we will ascertain delayed graft function (DGF) through center reports to UNOS. We will ascertain allograft failure through center reports to UNOS and new episodes of wait-listing and re-transplant collected by UNOS, Recipient mortality will be ascertained through the center reports to UNOS/SRTR and through the Social Security Death Master File.
4. Detailed Recipient Cohort

   A subset of over 1100 recipients of the Overall Cohort who had transplantation at any of our collaborating transplant centers will comprise this cohort. For the Detailed Subcohort, on-site coordinators will perform manual chart review and abstract more extensive data about each recipient including dialysis indications post-transplant, comorbidities, and specific doses of immunosuppression. For the Detailed Subcohort, we will also collect data on clinical events for up to five years after transplantation, including acute rejection and estimated glomerular filtration rate at the time of transplantation and at months 1, 3, 6, 12, 18, 24, 30, 36, 48 and 60 months after transplant.
5. Novel biomarkers will be measured in urine and perfusate

ELIGIBILITY:
Inclusion Criteria:

* Donor Cohort: Appropriate informed consent for research according to OPO policies
* Recipient Cohorts: Any recipient of at least one kidney from a deceased donor enrolled by our participating OPOs

Exclusion Criteria:

• Donor Cohort: Lack of adequate biospecimen quantity or quality as per protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population from which our Deceased-Donor Cohort will be selected is all potential deceased organ donors located in the regions serviced by our participating organ procurement organizations (OPOs).
  The recipient cohorts will be defined by the deceased donors enrolled in the study, and thus, the study population for this group is all recipients of kidneys from deceased organ donors procured in the regions serviced by our participating OPOs.
Sampling Method: Probability Sample
Enrollment: 1679 (Actual)
Dates: Start 2010-05-01; Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Delayed Graft Function | Assessed within first week of receiving renal transplant
  Receipt of dialysis within the first seven days post renal transplant
Death-Censored Graft Failure (Overall Cohort) | median of 4 years of follow-up
  Requirement of chronic dialysis or retransplantation after renal transplant.

SECONDARY OUTCOMES:
Graft Function (detailed cohort) | median of 4 years of follow-up
  Serum creatinine and estimated glomerular filtration rate at specified time points over a five year period.

CONTACTS AND LOCATIONS:
Overall Officials: Chirag R Parikh, MD PhD, Principal Investigator — Yale University
Locations (17):
- United States (17):
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Maryland Medical Center, Baltimore, Maryland
  - New England Organ Bank, Waltham, Massachusetts
  - Gift of Life Michigan, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - St. Barnabas Medical Center, Livingston, New Jersey
  - New Jersey Sharing Network, New Providence, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Organ Donor Network, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - NewYork-Presbyterian/ Columbia University Irving Medical Center, New York, New York
  - The New York Hospital (Cornell), New York, New York
  - Montefiore Medical Center, New York, New York
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Gift of Life Donor Program- Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Hall IE, Bhangoo RS, Reese PP, Doshi MD, Weng FL, Hong K, Lin H, Han G, Hasz RD, Goldstein MJ, Schroppel B, Parikh CR. Glutathione S-transferase iso-enzymes in perfusate from pumped kidneys are associated with delayed graft function. Am J Transplant. 2014 Apr;14(4):886-96. doi: 10.1111/ajt.12635. Epub 2014 Feb 24. PMID 24612768
- [Result] Hall IE, Reese PP, Weng FL, Schroppel B, Doshi MD, Hasz RD, Reitsma W, Goldstein MJ, Hong K, Parikh CR. Preimplant histologic acute tubular necrosis and allograft outcomes. Clin J Am Soc Nephrol. 2014 Mar;9(3):573-82. doi: 10.2215/CJN.08270813. Epub 2014 Feb 20. PMID 24558049
- [Result] Liu C, Hall IE, Mansour S, Thiessen Philbrook HR, Jia Y, Parikh CR. Association of Deceased Donor Acute Kidney Injury With Recipient Graft Survival. JAMA Netw Open. 2020 Jan 3;3(1):e1918634. doi: 10.1001/jamanetworkopen.2019.18634. PMID 31913491
- [Result] Puthumana J, Hall IE, Reese PP, Schroppel B, Weng FL, Thiessen-Philbrook H, Doshi MD, Rao V, Lee CG, Elias JA, Cantley LG, Parikh CR. YKL-40 Associates with Renal Recovery in Deceased Donor Kidney Transplantation. J Am Soc Nephrol. 2017 Feb;28(2):661-670. doi: 10.1681/ASN.2016010091. Epub 2016 Jul 22. PMID 27451287
- [Derived] Yaffe HC, von Ahrens D, Urioste A, Mas VR, Akalin E. Impact of Deceased-donor Acute Kidney Injury on Kidney Transplantation. Transplantation. 2024 Jun 1;108(6):1283-1295. doi: 10.1097/TP.0000000000004848. Epub 2023 Nov 22. PMID 37990359
- See also: Pubmed Link for Deceased Donor Study — https://www.ncbi.nlm.nih.gov/pubmed/?term=deceased+donor+study%2C+parikh+cr